CLINICAL TRIAL: NCT05457010
Title: Master Protocol for the Phase 1 Study of Cell Therapies for the Treatment of Patients With Relapsed or Refractory Acute Myeloid Leukemia or High-risk Myelodysplastic Syndrome, Including Long-term Safety Follow-up
Brief Title: Phase I Study of Cell Therapies for the Treatment of Patients With Relapsed or Refractory AML or High-risk MDS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arcellx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-201
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Arcellx; ARC-T cells; SparX; SPRX002; ACLX-002
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD123-Specific Adapter (SPRX002) and Universal CAR-Modified T Cell (ARC-T Cells) (Experimental): Arm 1: Phase 1 Study of monovalent CD123-Specific Adapter (SPRX002) and Universal CAR-Modified T cell (ARC-T Cells) for the Treatment of Patients with Relapsed or Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes
  Interventions: Biological: SPRX002; Biological: ARC-T Cells

INTERVENTIONS:
Biological: SPRX002 — SPRX002 is a soluble protein with a "TAG" region to which ARC-T cells bind and a binding region targeting CD123
Biological: ARC-T Cells — ARC-T Cells is a genetically modified autologous T-cell product. The T cell has a binding domain chimeric antigen receptor (CAR), which specifically binds to the "TAG" protein of the soluble protein antigen-receptor x-linker (sparX; specifically, SPRX002). When ARC-T cells bind to a "TAG" and the SPRX protein is bound to its target (in this case CD123), ARC-T cells are capable of activation, expansion, and killing (based on preclinical experiments).

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary activity of ARC-T cells and SPRX002 in participants with relapsed or refractory acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS)

DETAILED DESCRIPTION:
This is a Phase I open-label, safety, and dose-escalation study of ARC-T cells and SPRX002 in participants with relapsed or refractory AML or high-risk MDS. The study will have the following sequential phases: screening, enrollment, pretreatment with lymphodepletion (LD) chemotherapy, treatment with SPRX002 and ARCT cells, treatment extension with SPRX002, follow up, and long-term safety follow-up.

Following a single infusion of SPRX002 and ARC T (Day 0) and followed by regular administration of SPRX002 at the assigned dose level, both safety and efficacy data will be assessed. Dose limiting toxicities (DLTs) will be assessed through Day 28 and safety data will be collected throughout the study. Long-term safety data will be collected for up to 15 years per health authority guidelines. Efficacy will be assessed monthly for the first 6 months, then quarterly up to 2 years, or upon subject relapse.

ARC-T cells are a genetically modified autologous T-cell product. The T cell has been transduced using a third-generation lentiviral vector encoding a binding domain (referred to as AF101) chimeric antigen receptor (CAR), followed by CD8 spacer and transmembrane region that is fused to the intracellular signaling domains 4-1BB and CD3ζ. AF101 specifically binds to the "TAG" protein (referred to as Q26) of the soluble protein antigen-receptor x-linker (sparX; specifically, SPRX002).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. For AML Subjects: WHO-confirmed AML, other than APL, with no standard treatment options available (WHO AML Criteria 2016)

   a. Relapsed or refractory disease after at least 1 line of therapy, as defined by the following: i. Relapsed: Bone marrow blasts ≥5% following achievement of CR/Cri/MLFS

ii. Refractory: Failure to achieve CR/Cri/MLFS with evidence of persistent leukemia by blood and/or bone marrow examination after any of the following:

1. Failure on at least 1 cycle of an anthracycline-based induction therapy
2. At least 1 cycle of high or intermediate dose cytarabine containing induction regimen
3. At least 2 cycles of VEN-based lower intensity therapy, e.g., with HMA, or LDAC or cladribine+LDAC
4. At least 4 cycles of HMA-based therapy without venetoclax

3.For MDS Subjects: A diagnosis of MDS and ≥10% bone marrow blasts with indication of high-risk disease defined as those having resistant or refractory disease to at least one course of therapy including hypomethylating agents (e.g., decitabine or 5-azacitidine) given at conventional dose, schedule, and duration (e.g., cycle every 28 days and for at least 4 cycles) with or without venetoclax or other agents. Failure is defined as failure to attain a response, or relapse after prior response to HMA therapy per the modified IWG criteria.

4. Patients relapsing after allogeneic hematopoietic stem cell transplant (HSCT) >3 months prior are eligible if they have recovered from all transplant-related toxicities and are off all immunosuppression for at least 6 weeks.

5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1

6. Adequate organ function, including renal and hepatic function based on last clinical assessment performed within the screening period

1. Creatinine clearance ≥50 ml/min (Cockcroft-Gault or 24-hour urine collection in cases in which Cockroft-Gault is unreliable or if preferred by physician) and not on dialysis
2. Alanine aminotransferase <3 x upper limit of normal (ULN)
3. Aspartate aminotransferase <3 x the upper limit of normal (ULN)
4. Total bilirubin <2 x upper limit of normal (ULN) (except for patients with known or suspected history of Gilbert's Syndrome where up to 3x ULN is allowed)
5. Left Ventricular Ejection Fraction (LVEF) ≥45% by echocardiography (ECHO) or multi-gated acquisition (MUGA) scan
6. Pulse oxygenation ≥92% on room air
7. Prothrombin time test (PTT), prothrombin time (PT)/international normalized ratio (INR) <1.5 x ULN, unless on a stable dose of anti-coagulant for thromboembolic event (patients with any history of thromboembolic stroke; or history or Grade 2 (G2) or greater hemorrhage within 60 days are excluded)

   7. Resolution of adverse events (AEs) from any prior systemic anticancer therapy, radiotherapy, or surgery to Grade 1 or baseline (except G2 alopecia and G2 sensory neuropathy)

   8. Prior allogeneic stem cell transplant is allowed, provided the subject has recovered from all AEs, there is no ongoing graft-versus-host-disease (GvHD) and subject is not on taking any immunosuppressive medications to prevent GvHD

   9. Male and females of childbearing potential must agree to use highly effective methods of birth control through 6 months after the dose of study treatment.

   10. Patients must have an identified potential donor and transplant strategy/plan prior to initiation of the lymphodepletion regimen to ensure availability of hematopoeitic stem cells (HSCs) for potential urgent allogeneic HSC transplant (HSCT) if needed for persistent bone marrow aplasia without evidence of residual leukemia. Transplant decision making would be a discussion between subject and investigator due to potential for treatment-related mortality and is not required

   11. Willing to comply with and able to tolerate study procedures, including Long-Term Safety Follow-up lasting up to 15 years

   12. Life expectancy > 3 months

   13. Subject's apheresis product from non-mobilized cells is received and accepted for cell processing by manufacturing site. NOTE: apheresis will be accepted only after all other eligibility criteria have been met

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia (APL) or EMD-only disease
2. Patients with active CNS involvement. Subjects may be cleared of CNS involvement if there has been no evidence of CNS involvement for at least 3 months prior to enrollment. For instance, CSF samples showing no evidence of blasts by CSF cytology, no clinical signs or symptoms, or no radiological findings concerning for CNS involvement.
3. Hyperleukocytosis (≥25,000 blasts/μL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy. (Note: Subjects may be receiving or may receive hydroxyurea to maintain or control hyperleukocytosis)
4. Previous treatment with an investigational gene or chimeric antigen receptor therapy (Note: May be permitted after discussion with Medical Monitor)
5. Previous treatment with a CD123 directed therapy (T-cell engager or ADC)
6. Use of any anti-AML/MDS directed chemotherapy or targeted therapy (except hydroxyurea therapy) or immunosuppressive agents (physiologic doses are allowed), within 14 days or 5 half-lives (whichever is shorter) prior to the date of leukapheresis and use of any anti-AML/MDS directed monoclonal antibody within 28 days prior to date of leukapheresis
7. Known infection with Human Immunodeficiency Virus or Human T-Cell leukemia/lymphoma virus type 1 (HTLV-1)
8. A known hypersensitivity or severe allergy to study drug components including dimethyl sulphoxide (DMSO) and human serum albumin
9. Contraindication to cyclophosphamide or fludarabine
10. Subject has systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate treatment (Note: Isolated fever may not constitute active infection in and of itself, (e.g., related to disease)
11. Severe uncontrolled intercurrent illness including:

    1. Cardiovascular disease
    2. Symptomatic congestive heart failure
    3. Unstable angina, arrythmia, or myocardial infarction (MI) within 6 months prior to screening
    4. Significant pulmonary dysfunction
    5. Uncontrolled thromboembolic events or recent severe hemorrhage
    6. Any history of pulmonary embolism (PE) ever or deep vein thrombosis (DVT) within 3 months of screening. Therapeutic dosing of anticoagulants (e.g., warfarin, low molecular weight heparin, Factor Xa inhibitors) is allowed for history of DVT if greater than 3 months from time of screening) Note: Central line thrombosis not requiring anticoagulation will not be excluded and will not require a 3-month screening window
    7. Autoimmune disease
12. Seropositive for and with evidence of active hepatitis B or C infection at time of Screening

    1. Subjects with a history of hepatitis B but have received antiviral therapy and have non-detectable viral DNA for 6 months are eligible
    2. Subjects seropositive because of hepatitis B virus vaccine with no signs or active infection are eligible
    3. Subjects who had hepatitis C but have received antiviral therapy and show no detectable hepatitis C virus (HCV) viral RNA for 6 months are eligible
13. Any sign of active CNS pathology within 6 months of screening including history of epilepsy, seizure requiring anti-seizure medications, paresis, aphasia, stroke, severe brain injury, dementia, cerebellar disease, Parkinson's disease, organic brain syndrome or psychosis. Subarachnoid hemorrhage or central nervous system (CNS) bleed within 3 months of screening
14. Subject has active malignant tumors other than AML/MDS that requires active antineoplastic or radiation therapy at the time of screening. Maintenance therapy or hormonal therapy for well-controlled malignancy is allowed
15. Females who are pregnant or breastfeeding
16. Subjects with any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in study (or full access to medical records) as written including follow up, the interpretation of data or place the subject at unacceptable risk are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), including dose-limiting toxicities (DLTs) and establish recommended Phase II dose (RP2D) | 24 months
  The RP2D will be determined based on the totality of data, including the maximum tolerated dose (MTD); if applicable, and other endpoints such as observed efficacy, pharmacokinetics (PK), pharmacodynamics (PD), and other safety endpoints (adverse events (AEs), laboratory assessment, vital signs, and physical examinations)

SECONDARY OUTCOMES:
Anti-Tumor Activity | 24 months
  Serial blood and bone marrow sampling to determine response to treatment by modified International Working Group (IWG) Response Criteria in AML and MDS, or other appropriate response criteria for the malignancy under study, such as overall response rate, composite complete remission rate, and rate of negative minimum residual disease (MRD)
Pharmacokinetics (PK) | 24 months
  Quantification of ARC-T cells and SPRX002 using vector copy number (VCN) on peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Tim Welliver, MD, PhD, Study Chair — Arcellx, Inc.
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Montefiore Einstein Cancer Center, New Rochelle, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No